CLINICAL TRIAL: NCT06019845
Title: The MAGiC™ Cardiac Ablation Feasibility Study
Brief Title: The MAGiC™ Cardiac Ablation European Study
Acronym: MAGiC-FEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stereotaxis (Industry)
Collaborators: Osypka AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MFEAS-001; CIV-23-10-044301 (Other: EUDAMED)
Record Dates: First submitted 2023-08-23; First posted 2023-08-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Arrhythmias, Cardiac
Keywords: Atrial Fibrillation; Atrial Flutter; Ventricular Tachycardia; Supraventricular Tachycardia; Ablation; Premature Ventricular Contractions
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Tachycardia, Ventricular; Tachycardia, Supraventricular; Ventricular Premature Complexes | interventions — Magic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Magnetic Interventional Ablation Catheter (MAGiC™)
  Interventions: Device: MAGiC™

INTERVENTIONS:
Device: MAGiC™ — Robotic magnetic radiofrequency (RF) ablation catheter

SUMMARY:
The purpose of the first phase of this feasibility study is to gather safety and performance data on MAGiC to support European marketing approval.

DETAILED DESCRIPTION:
The purpose of the first phase of this feasibility study is to gather safety and performance data on MAGiC to support European marketing approval. After MAGiC obtains European approval, the study will be amended and expanded to collect Post-Market Clinical Follow-up data.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or older at time of consent);
* Eligible for ablation procedures of an atrial or ventricular arrhythmia per European Heart Rhythm Association (EHRA) guidelines, with at least one (1) documented episode of the tachyarrhythmia to be treated within the previous six (6) months;
* Able to be safely exposed to magnetic fields;
* Willing and capable to attend scheduled follow up visits at the investigational site for the study duration (up to 12 months)
* Willing and able to provide informed consent.

Exclusion Criteria:

* Unable to be safely exposed to magnetic fields due to Magnetic Resonance Imaging Unsafe device (implanted device or device that cannot be safely removed for the procedure)
* Unable to remain comfortable or hemodynamically stable in the supine position for an extended period of time
* Weight exceeding 200 kg (the weight limit of the table)
* For female patients of childbearing potential: pregnancy at the time of the procedure or unwilling to take a pregnancy test
* Presence of intracardiac thrombus at the time of the procedure
* Where MAGiC would need to cross a prosthetic valve
* Use of MAGiC in the coronary arteries
* A history of sensitivity to foreign objects or extreme allergies
* Acute illness or active systemic infection
* Histological or anatomical abnormalities that may lead to post-operative complications including diminished resistance to infection
* Hemodynamic instability
* Unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation
* Acute myocardial infarct (within the previous 30 days)
* Recent cardiac surgery (within the previous 60 days)
* Unstable angina
* History of embolism (cerebrovascular accident, transient ischemic attack, systemic embolism) in the previous 30 days
* Previous cardiac ablation within the previous 30 days
* Concomitant arrhythmia(s) requiring active treatment at this time or in the 90 days prior to enrollment (Day -90 to Day 0)
* Currently or in the 30 days prior to consent, participation in an interventional clinical trial
* Significant uncontrolled or unstable medical problems which, in the opinion of the Investigator, would preclude enrollment in and completion of the study (limitation on survival).
* Any reason or condition that, in the judgement of the investigator, makes the patient ineligible for the investigation.
* For Atrial Fibrillation only: persistent Atrial Fibrillation (continuous Atrial Fibrillation lasting longer than 7 days)
* For Atrial Fibrillation only: Presence of any device that would interfere with planned access: Patent Foramen Ovale occlusion/closure device, patch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Acute Performance | hospital discharge - up to 7 days post procedure
  The primary endpoint is to estimate the acute procedural success across a range of treated arrhythmias.
Acute Safety | hospital discharge - up to 7 days post procedure
  Freedom from major adverse events (MAE) related to MAGiC.

SECONDARY OUTCOMES:
Chronic Success | 3 months, 6 months, 12 months
  Percentage of subjects free from the treated index arrhythmia at the relevant chronic timepoint.
Safety Events | 3 months, 6 months, 12 months
  Rate of subjects experiencing investigational device-related adverse events and procedure-related adverse events.
Onset of Procedure-related New Arrhythmia | 3 months, 6 months, 12 months
  Percentage of subjects who experience the onset of a new arrhythmia related to the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Lowry, Study Director — Stereotaxis
Locations (2):
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- Vilniaus universiteto ligoninė Santaros klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No